CLINICAL TRIAL: NCT05622071
Title: A Multicentric National Phase II Trial Assessing TIslelizumab in Monotherapy for Patients With Hepatocellular Carcinoma Child-Pugh B and ALBI Grade 1 or 2 Liver Function Score
Brief Title: Testing Immunotherapy for Patients With Liver Cancer and Moderately Altered Liver Functions
Acronym: HESTIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-GIG-2003
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2024-09

CONDITIONS: Hepatocellular Carcinoma by BCLC Stage
Keywords: Hepatocellular Carcinoma; tislelizumab; monotherapy; Child-Pugh B; ALBI grade 1 or 2 liver function score
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: Multicentre, national, monotherapy, open-label, phase II single-arm study
Masking Description: Tislelizumab will be administered every 3 weeks IV for a maximum of 2 years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SINGLE ARM (Experimental): Tislelizumab 200 mg will be administered every 3 weeks IV. Treatment will be continued until progression or limiting toxicities, for a maximum duration of 2 years and with an average duration of 4 months
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200 mg will be administered every 3 weeks IV for a maximum of 2 years
  Other Names: BGB-A317

SUMMARY:
Liver cancer is the third leading cause of cancer-related deaths worldwide. The majority of primary liver cancers occur as hepatocellular carcinoma (HCC), the incidence of which is increasing in many parts of the world. The vast majority of HCC cases occur in the setting of liver cirrhosis, usually due to chronic viral infections with hepatitis C or hepatitis B, alcohol consumption, non-alcoholic fatty liver disease or diabetes. The degree of underlying liver disease, as well as the stage of the tumour and the general condition of the patients, should therefore be taken into account when deciding on the treatment of HCC. Most patients with HCC have advanced disease at the time of diagnosis, or have recurrent disease after potentially curative treatments.

Tislelizumab showed enhanced cellular functional activities by blocking PD-1-mediated reverse signal transduction and activating human T cells and primary peripheral blood mononuclear cells in vitro.

Based on this preliminary safety profile, and knowing that there is antitumour activity, we can offer tislelizumab as a single agent in patients with unresectable HCC.

HESTIA study is a multicentric French national phase II trial assessing tislelizumab in monotherapy for patients with Hepatocellular Carcinoma Child-Pugh B and ALBI grade 1 or 2 liver function score.

It is planned to include 50 patients in the study. All patients will be recruited in France. The study will be presented to eligible patients at participating centres and an information note will be provided. No advertising material is planned for this study.

To be eligible, patients must meet all the following criteria to be ≥18 years old, with histologically proven Hepatocellular Carcinoma (HCC), pre-treated or not with a tyrosine kinase inhibitor and Child-Pugh B cirrhosis, ALBI (Albumin-Bilirubin) grade 1 or 2 and BCLC (Barcelona Clinic Liver Cancer Group) B or C and with no more than 50% liver invasion of tumour disease.

DETAILED DESCRIPTION:
The primary objective is to assess efficacy of anti-PD1 (in terms of Objective Response Rate [ORR] based on Best Overall Response across all time-points as defined by RECIST v1.1) in the Child-Pugh B / ALBI grade 1/2 population.

Secondary objectives are :

* To assess safety of anti-PD-1
* To assess efficacy in terms of:

  * Objective Response Rate based on best overall response across all time-point according to mRECIST and iRECIST tumor response evaluation
  * Overall survival (OS)
  * Progression-free survival (PFS)
  * Time to progression (TTP)
* To assess Quality of Life according to EORTC QLQ-C30 and HCC-18.

In order to confirm the eligibility of patients, a clinical examination, biological blood tests, ECG, CT scan and a urine or blood pregnancy test for women of childbearing age will be performed. A quality of life questionnaire will be administered to patients. Patients will also be asked to agree to a full eye examination by an ophthalmologist prior to the start of treatment to determine that there is no risk of worsening the patient's visual acuity with treatment with tislelizumab.

After enrolment in the study, the patient will be required to visit the hospital every 3 weeks to receive intravenous treatment for up to 2 years.

Once the treatment is completed, the patient will be seen at follow-up visits for 2 years, initially every 3 months for the first year and then every 6 months for the second year.

Assessment of tumour response by CT or MRI will be done after the start of treatment at weeks 9, 18, 27, 54 and every 12 weeks until disease progression and throughout the treatment period. Tumour assessment by CT or MRI will be performed 2 years after the start of treatment or upon disease progression.

Patients will be asked to consent to the use of a collected tumour sample, as well as to the collection of blood samples, for future scientific research which includes, but is not limited to, the detection of DNA, RNA and protein biomarkers.

An independent Study Monitoring Board (DSMB), with expertise and experience in the pathology, and without direct involvement in the conduct of the study, will be set up specifically to ensure optimal safety monitoring during the early phase of the study and the feasibility of at least 2 treatment injections (6 weeks from inclusion), an early stopping rule has been defined for the first 20 patients included. This method was chosen for the evaluation of serious adverse events (SAEs), which may occur relatively early in this trial. A high frequency of occurrence may necessitate early termination of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Patient presenting with histologically-proven Hepatocellular Carcinoma (HCC), or HCC defined by typical imaging findings (EASL criteria), if no biopsy could be performed safely
3. Pretreated or not by tyrosine kinase inhibitors (e.g., sorafenib, lenvatinib, regorafenib, cabozantinib)
4. Child-Pugh B cirrhosis
5. ALBI (Albumin-Bilirubin) grade 1 or 2
6. BCLC (Barcelona Clinic Liver Cancer Group) B or C
7. Availability of biopsy specimen at study enrolment (taken within 3 months of enrolment with the exception of cases where biopsy could not be performed safely)
8. ECOG Performance status ≤2
9. Adequate organ function as indicated by the following laboratory values:

   1. Patients must not have required a blood transfusion or growth factor support ≤14 days before sample collection at screening for the following:

      * Absolute neutrophil count (ANC) ≥1.5 x 10⁹/L
      * Platelets ≥75 x 10⁹/L
      * Hemoglobin ≥90 g/L
   2. Serum creatinine ≤1.5 x upper limit of normal (ULN) or estimated Glomerular Filtration Rate ≥60 mL/min/1.73 m²
   3. Serum total bilirubin ≤3 mg/dL
   4. Liver function: ASAT and ALAT ≤5 ULN, albumin >2.0 g/dL
10. Presence of measurable and evaluable disease according to RECIST v1.1
11. Women of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study, and ≥120 days after the last dose of tislelizumab, and have a negative urine or serum pregnancy test ≤7 days of first dose of study drug. In case of a urine pregnancy test, it must be a highly sensitive urine pregnancy test
12. Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study and for ≥120 days after the last dose of tislelizumab. A sterile male is defined as one for whom azoospermia has been previously demonstrated in a semen sample examination as definitive evidence of infertility. Males with known "low sperm counts" (consistent with "sub-fertility") are not to be considered sterile for purposes of this study
13. Patients must have provided consent for the study by signing and dating a written informed consent form prior to any study specific procedures, sampling, or analyses. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent
14. Patient consent to the use of their collected tumour specimen, as well as blood samples as detailed in the protocol for future scientific research which includes but not limited to DNA, RNA, and proteinbased biomarker detection
15. Patient affiliated to a social security regimen
16. Men and women patients must consent to not donate or bank sperm or ova during treatment and for 120 days after treatment stop

Exclusion Criteria:

1. More than 50% of the liver is affected by the HCC (according to investigators evaluation)
2. Fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
3. Previous treatment with immunotherapy (anti-PD-1, anti-PD-L1, or anti-CTLA-4 agents)
4. History of active autoimmune disease. Note: Patients with the following diseases are not excluded and may proceed to further screening:

   1. Type I diabetes
   2. Hypothyroidism (provided it is managed with hormone replacement therapy only)
   3. Controlled celiac disease
   4. Skin diseases not requiring systemic treatment (e.g., vitiligo, psoriasis, alopecia)
   5. Any other disease that is not expected to recur in the absence of external triggering factors
5. History of interstitial lung disease, non-infectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases
6. Any of the following cardiovascular risk factors:

   1. Cardiac chest pain, defined as moderate pain that limits instrumental activities of daily living, ≤28 days before first dose of study drug
   2. Pulmonary embolism ≤28 days before first dose of study drug
   3. Any history of acute myocardial infarction ≤6 months before first dose of study drug
   4. Any history of heart failure meeting New York Heart Association (NYHA) Classification III or IV ≤6 months before first dose of study drug
   5. Any event of ventricular arrhythmia ≥ Grade 2 in severity ≤6 months before first dose of study drug
   6. Any history of cerebrovascular accident ≤ 6 months before first dose of study drug
   7. Uncontrolled hypertension: systolic pressure ≥160 mmHg or diastolic pressure ≥100 mmHg despite anti-hypertension medications before first dose of drug
   8. Any episode of syncope or seizure before first dose of study drug
7. Patients with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers whose HBV DNA is >500 IU/mL or patients with active hepatitis C virus (HCV) should be excluded. Note: Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B (HBV DNA <500 IU/mL), and cured hepatitis C patients can be enrolled
8. Known primary immunodeficiency or active HIV
9. Immunosuppression, including subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg/day prednisone equivalent) ≤14 days before inclusion. Note: Patients who are currently or have previously been on any of the following steroid regimens are not excluded:

   1. Adrenal replacement steroid (dose ≤10 mg daily of prednisone or equivalent)
   2. Topical, ocular, intra-articular, intranasal, or inhaled corticosteroid with minimal systemic absorption
   3. Short course (≤7 days) of corticosteroid prescribed prophylactically (e.g., for contrast dye allergy) or for the treatment of a non-autoimmune condition (e.g., delayed-type hypersensitivity reaction caused by contact allergen)
10. Live vaccine within 4 weeks of first dose of study drug. Note: Seasonal vaccines for influenza are generally inactivated vaccines and Covid vaccination with non-live vaccine are allowed. Intranasal vaccines are live vaccines, and are not allowed
11. Transplanted liver, or patient with intent for transplantation
12. Received locoregional therapy to the liver (TACE, transcatheter embolization, hepatic arterial infusion, radiation, radioembolization or ablation) in the 4 weeks before inclusion
13. Prior malignancy active within the previous 3 years of inclusion except for locally curable cancers considered cured or successfully resected, such as basal or squamous cell skin cancers, superficial bladder cancer, or gastric cancers, or carcinoma in situ of the prostate, cervix, or breast carcinomas. Any oncological concomitant treatment are not allowed during the treatment period
14. Has received any herbal medicine used to control cancer with immunostimulant properties that may interfere with liver function within 14 days of the first study drug administration
15. Pregnant woman or breast-feeding women or patient with no adequate contraception
16. Participation in another therapeutic trial within the 30 days prior to study inclusion
17. Patients deprived of their liberty or under protective custody or guardianship
18. Patients unable to adhere to the protocol for geographical, social, or psychological reasons
19. Patients eligible for treatment by TACE or SIRT are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 48 months
  Objective response rate (ORR) is the percentage of patients with a best response during treatment being either complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Frequency of limiting toxicity | From inclusion, up to 6 months
  Frequency of limiting toxicity is defined as any adverse event related to the experimental drug, and leading to definitive treatment discontinuation according to the investigator, before the second injection.
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
Frequency of related and not related adverse events | From inclusion, up to 48 months
  Frequency of all adverse events occurring during the treatment period and until 3 months after treatment discontinuation.
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
Overall survival | From inclusion to death from any cause, up to 52 months
  The overall survival (OS) is the length of time from randomization that patients enrolled in the study are still alive.
Progression-free survival | From inclusion to disease progression or death, up to 52 months
  The progression-free survival (PFS) is the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse.
Time to progression | From inclusion to radiographic disease progression, up to 52 months
  Time to progression is the length of time patients leave without radiological disease progression.
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, every 6 week for 1 year, then every 4 months, up to 52 months
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of life questionnaire - Hepatocellular Carcinoma (QLQ-HCC-18) | At baseline, every 6 week for 1 year, then every 4 months, up to 52 months
  This EORTC hepatocellular carcinoma specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-HCC18 contains 18 items to assess symptoms hepatocellular-related symptoms. These items are grouped into 6 domains: fatigue, body image, jaundice, nutrition, pain, and fever. Two single items address abdominal swelling and sex life. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale; a higher score represents a more severe symptom or problem.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Edeline, MD PhD, Principal Investigator — CLCC UNICANCER EUGENE MARQUIS
Locations (10):
- France (10):
  - CHU Angers, Angers
  - Hôpital Avicenne, Bobigny
  - CHU Beaujon, Clichy
  - Hôpital Michallon, Grenoble
  - CHU La Croix Rousse, Lyon
  - Hôpital Saint Joseph, Marseille
  - Institut Paoli Calmette, Marseille
  - CHU Saint Eloi, Montpellier
  - Centre Eugene Marquis, Rennes
  - CHRU Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edeline J, Blanc JF. Difficulties for providing evidence in hepatocellular carcinoma with Child-Pugh B liver function. Liver Int. 2023 Feb;43(2):274-275. doi: 10.1111/liv.15495. No abstract available. PMID 36680319